CLINICAL TRIAL: NCT01896180
Title: A Pilot, Single-Masked Study to Compare the Safety and Efficacy of ALZ-1101 (Latanoprost 0.005%/Dorzolamide 2.0%) to Latanoprost Ophthalmic Solution, 0.005% in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension With Intraocular Pressure Inadequately Controlled By Latanoprost
Brief Title: Study to Compare the Safety and Efficacy of ALZ-1101 to Latanoprost in Patients With Intraocular Pressure Inadequately Controlled by Latanoprost
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alleanza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALZ-1101-101
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension; Elevated Intraocular Pressure
Keywords: POAG; OHT; OHTN; IOP
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALZ-1101 (Experimental): ALZ-1101 ophthalmic solution dosed as 1 drop, once daily in the evening via topical ocular adminstration
  Interventions: Drug: ALZ-1101
- Latanoprost (Active Comparator): Latanoprost 0.005% ophthalmic solution dosed as 1 drop, once daily in the evening via topical ocular administration
  Interventions: Drug: Latanoprost

INTERVENTIONS:
Drug: ALZ-1101 — ALZ-1101 Ophthalmic Solution
  Arms: ALZ-1101
Drug: Latanoprost — Latanoprost 0.005% Ophthalmic Solution
  Arms: Latanoprost

SUMMARY:
This is a pilot, proof of concept study to evaluate the safety and efficacy of ALZ-1101 dosed once daily for 28 days compared to latanoprost 0.005% ophthalmic solution in patients with elevated intraocular pressure not adequately controlled with latanoprost.

DETAILED DESCRIPTION:
This is an exploratory, pilot, proof of concept Phase 2 study. The objectives include the comparison of efficacy of ALZ-1101 to latanoprost 0.005% ophthalmic solution in reducing elevated intraocular pressure (IOP) in patients with primary open angle glaucoma or ocular hypertension who have IOP not adequately controlled with latanoprost.

70 Subjects (35 per arm) will be treated once daily (QD) in the evening with either ALZ-1101 or latanoprost for 28 days.

Efficacy will be assessed at 3 separate times (8 AM, 10 AM and 4 PM) on each treatment visit (Days 0, 7, 14 and 28) by Goldmann applanation tonometry.

Safety assessments will include slit lamp examination/anterior chamber cell and flare grading, ophthalmoscopy/fundus examination, visual acuity, visual field testing and colelction of adverse events. Subject rating of study medication comfort will be collected at each visit.

Primary efficacy endpoint is the between-group comparison of the mean IOP at the 10 am time point at visit 5 (Day 28). Secondary endpoints include the between-group comparisons of the mean change from baseline in IOP at all time-points, between group comparison of the mean change from baseline in diurnal IOP at all post-baseline visits and the proportion of subjects with IOP ≤ 18 mm Hg at all time points at all post-baseline visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Primary open-angle glaucoma or OH on treatment with latanoprost 0.005% QD.
3. At least one eye with IOP > 18 mm Hg but ≤ 28 mm Hg at all time points (8 AM, 10 AM, and 4 PM) while on latanoprost monotherapy QD at Screening and Baseline (Day 0) visits. Measurements will be taken each visit at 8 AM, 10 AM, and 4 PM (each ± 30 minutes), with AM measurements of IOP at least 2 hours apart. Screening must be at least one week before but within 2 weeks prior to Baseline.
4. On latanoprost 0.005% QD for at least 4 weeks prior to randomization.
5. Shaffer gonioscopic grade of ≥ 3 (in at least 3 quadrants) in both eyes.
6. Stable corrected Snellen visual acuity (VA) better than 20/200 in the study eye.
7. Central corneal thickness between 480-620 μm in the study eye.
8. Female subjects must be 1-year postmenopausal, surgically sterilized, or women of childbearing potential with a negative urine pregnancy test at Visit 1. Women of childbearing potential must use an acceptable form of contraception throughout the study. Acceptable methods include the use of at least one of the following: intrauterine (intrauterine device), hormonal (oral, injection, patch, implant, ring), barrier with spermicide (condom, diaphragm), or abstinence.
9. Provide signed written consent prior to participation in any study-related procedures.

Exclusion Criteria:

1. A mean deviation of < -20 dB on visual field (VF) assessment.
2. Presence of a scotoma within 5°of fixation on VF.
3. Aphakia.
4. Use of any antiglaucoma medication in addition to latanoprost QD within 2 weeks prior to Visit 1 or during the study period.
5. Use of any topical ophthalmic steroid or nonsteroidal anti-inflammatory drug (NSAID) within 2 weeks prior to Visit 1 or during the study period.
6. Use of systemic carbonic anhydrase inhibitor within 2 weeks prior to Visit 1 or during the study period.
7. Ocular surgery or ocular laser treatment of any kind within 3 months prior to Visit 1 or during the study period.
8. Any history of glaucoma surgery (laser or non-laser).
9. History of ocular allergy/inflammation and/or severe blepharitis and/or uveitis. Seasonal allergic conjunctivitis is acceptable (avoid enrollment of subjects who may experience seasonal flare-up during the study period). Mild blepharitis/blepharoconjunctivitis, typically associated with prostaglandin usage, is acceptable.
10. History of ocular trauma or ocular infection within 3 months of Visit 1.
11. History of herpes simplex keratitis.
12. Current proliferative diabetic retinopathy or age-related macular degeneration, unless deemed not clinically significant by the Investigator.
13. Severe dry eye (eg, clinically relevant superficial punctate keratitis, epithelial erosions of the cornea, and/or use of dry eye medication [including artificial tears] with a frequency exceeding 8 applications per day).
14. Contact lens wear within one week prior to Visit 1 or during the study period (contact lens wear in an untreated fellow eye is allowed).
15. Angle closure or occludable angles (Shaffer gonioscopic grade of < 3).
16. Cataract that compromises visualization of the fundus.
17. Cup-to-disc (C/D) ratio of > 0.8.
18. Any secondary glaucoma or OH (eg, congenital glaucoma, closed-angle glaucoma, uveitic glaucoma, or pseudoexfoliation syndrome).
19. Pregnancy or lactation.
20. Uncontrolled asthma (defined as asthma that does not respond to the maximum guideline directed therapy).
21. Allergy to prostaglandin analogues or carbonic anhydrase inhibitors.
22. Allergy to benzalkonium chloride.
23. History of moderate or severe renal or hepatic impairment.
24. Participation in any study of an investigational product within 30 days prior to Visit 1 or at any time during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Goldmann applanation tonometry | 28 days
  Between-group comparison of the mean IOP values at the 10 AM time point at Visit 5 (Day 28).

SECONDARY OUTCOMES:
Goldmann applanation tonometry | 28 days
  Between-group comparison of the mean change from baseline in IOP at all time points at all post-baseline visits
Goldmann applanation tonometry | 28 days
  Between-group comparison of the mean change from baseline in diurnal IOP at all post baseline visits
Goldmann applanation tonometry | 28 days
  The proportion of subjects with IOP ≤ 18 mm Hg at all time points at all post-baseline visits
Safety | 28 days
  Assessment of the safety and tolerability will be assessed by slit lamp examination/anterior chamber cell and flare grading, ophthalmoscopy (cup-to-disc ratio)/dilated fundus examination, corrected Snellen visual acuity, VF testing, and adverse event assessment. Comfort data (subjective) will also be collected at each visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Morrow, Georgia, United States